CLINICAL TRIAL: NCT06477367
Title: The Effect of Video-Based Breathing Exercises Taught to COPD Patients on Dyspnea Severity, Activity Level, and Sleep Quality
Brief Title: Changes in Dyspnea, Activity and Sleep in COPD by Video-Based Breathing Exercises
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Ayfer Bayındır Çevik, Assc. Prof, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BartınU_Bayındır Cevik_001
Record Dates: First submitted 2024-06-04; First posted 2024-06-27 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; patient with COPD; pursed lip breathing exercise; video-based breathing exercises; dyspnea; sleep quality; activity level; diaphragmatic breathing exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group receiving video-based training (Experimental): Researchers will present a 5-7 minute instructional video aimed at helping participants recall the technique for performing the exercises. These instructional videos will be sent to the researchers' mobile phones via WhatsApp. Participants will be instructed to perform the exercises three times a day for 15 minutes each, for a period of 30 days. To encourage regular exercise, participants will be provided with an exercise diary, and researchers will send reminder SMS messages at the same time every day.
  Interventions: Other: Video-Based Breathing Exercises
- The group not receiving video-based training (No Intervention): The control group will receive the clinic's routine dyspnea care protocol. After thirty days, final tests will be administered to both groups, and the research will be concluded.

INTERVENTIONS:
Other: Video-Based Breathing Exercises — Researchers will present a 5-7 minute instructional video aimed at helping participants recall the technique for performing the exercises. These instructional videos will be sent to the researchers' mobile phones via WhatsApp. Participants will be instructed to perform the exercises three times a day for 15 minutes each, for a period of 30 days. To encourage regular exercise, participants will be provided with an exercise diary, and researchers will send reminder SMS messages at the same time every day. The control group will receive the clinic's routine dyspnea care protocol. After thirty days, final tests will be administered to both groups, and the research will be concluded.
  Arms: The group receiving video-based training

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is one of the most prevalent and high-mortality chronic diseases worldwide. Symptoms such as dyspnea, cough, sleep disturbances, fatigue, restricted activity levels, anxiety, and depression develop in COPD patients, negatively affecting their quality of life. Dyspnea, associated with various symptoms in COPD patients such as reduced activity levels and sleep disturbances, is a significant issue. Therefore, effective management of dyspnea will contribute to reducing other important problems associated with COPD.

One of the non-pharmacological methods used in managing these symptoms associated with COPD is breathing exercises. Particularly, pursed-lip breathing exercises and diaphragmatic breathing exercises are recommended for symptom management in COPD patients in the literature.

The aim of this study was to learn the effects of video-based breathing exercises (pursed lips and diaphragmatic breathing) training given to COPD patients over 18 years of age on the severity of dyspnea experienced by the patient, activity level and sleep quality. The main question it aims to answer is:

Does the use of video-based breathing exercises for 30 days result in a decrease in dyspnea severity and an increase in activity level and sleep quality in COPD patients over 18 years of age? Patients will receive video-based breathing exercises lasting approximately 5-7 minutes and will perform the breathing exercises regularly for 30 days, keep a diary and receive follow-up messages (sms). Afterwards, dyspnea severity, activity level and sleep quality will be assessed again, both in the group itself and in comparison with the control group that did not receive this education and follow-up.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) stands as a prominent progressive chronic condition, with approximately 210 million individuals affected globally, placing it third in terms of global mortality. COPD is recognized as a widespread, preventable, and manageable ailment marked by ongoing airflow restriction linked to chronic inflammation triggered by harmful gases and particles. Patients with COPD commonly experience symptoms like shortness of breath, coughing, disrupted sleep, fatigue, limited physical activity, as well as feelings of anxiety and depression.

Nurses play a crucial role in evaluating and addressing symptoms in COPD patients. They can utilize non-pharmacological techniques such as respiratory exercises, progressive relaxation exercises, reflexology, and yoga to help manage and alleviate dyspnea. Pursed-lip breathing, deep breathing, and diaphragmatic breathing exercises are commonly recommended for controlling hyperventilation and addressing dyspnea in COPD patients. Pursed-lip breathing has been shown to lower respiratory rate, decrease carbon dioxide levels, and increase oxygen levels and tidal volume in COPD patients. Additionally, diaphragmatic breathing exercises have been found to boost tidal volume and oxygen levels while reducing respiratory rate in COPD patients.

Sleep problems develop in 40% of COPD patients. Dyspnea in COPD patients often leads to sleep disturbances. Additionally, cough and sputum-induced insomnia affect daily life activities in COPD patients. Adequate sleep has a positive effect on respiratory and gas exchange functions in respiratory system diseases. Therefore, managing dyspnea in COPD patients will also reduce their sleep problems.

Physical activity level is associated with mortality in COPD patients. Furthermore, it has been reported that good physical activity reduces the severity of COPD-related symptoms and improves quality of life. Factors such as dyspnea, lung capacity, and inflammation negatively affect activity levels in COPD patients. Studies in the literature suggest that physical exercise programs rather than respiratory exercises increase physical activity levels in COPD patients.

In conclusion, while studies in the literature report positive effects of respiratory exercises on dyspnea management, no studies examining the effect of respiratory exercises on sleep quality and physical activity were found. This study is planned to investigate the effect of pursed-lip breathing exercises and diaphragmatic breathing exercises on dyspnea severity, activity level, and sleep quality in COPD patients.

Research Method:

The study is planned as a randomized controlled design.

Data Collection Tools:

* 6-minute walk test:This test is used to evaluate functional capacity by measuring the distance walked within a certain period of time. In the 6-minute walk test, the patient walks as fast as possible, but without running, in a straight corridor of 30 meters. The distance walked is measured. During the test, the patient should not change their pace or speed. It is known that patients with poor 6-minute walk test results have a poor prognosis.
* Patient Information Form: In the form created in line with the literature information; socio-demographic information of the participant, information about the disease and other chronic diseases, medications used, and habits are obtained.
* Modified Borg Scale (MBS)
* Saint George Respiratory Questionnaire (SGRQ)
* Asthma and COPD Sleep Scale

Data Collection:

Patients receiving treatment for COPD at Bartın State Hospital Chest Diseases Service will form the sample. Patients who meet the inclusion criteria for the study will be randomized using a computer-assisted randomization system. Informed Voluntary Consent Form will be obtained from patients who agree to participate in the study, and then the Patient Information Form, Modified Borg Scale, Saint George Respiratory Questionnaire (Activity sub-score), and Asthma and Chronic Obstructive Pulmonary Disease Sleep Scale will be completed. After the pre-test, patients in the experimental group will be taught the pursed-lip breathing exercise and diaphragmatic breathing exercise recommended for COPD patients by the Turkish Thoracic Society. Additionally, patients will be shown a 5-7 minute instructional video prepared by the researchers regarding this. The educational videos will be sent to the researchers' mobile phones via WhatsApp for patients to remember the exercise technique. Patients will be instructed to perform these exercises regularly for 15 minutes three times a day for four weeks. To ensure that patients perform the exercises regularly, an exercise diary will be created and provided to them, and a reminder SMS message will be sent by the researchers at the same time every day. The control group will receive the clinic's routine dyspnea care protocol. After four weeks, final tests will be administered to both groups, and the study will be concluded.

Population and Sample:

The population of the study consists of patients treated with COPD diagnosis at Bartın State Hospital Chest Diseases Service. The sample size was calculated as 56 patients, with 28 in the intervention group and 28 in the control group, taking into account data obtained from a similar study with d=0.68, power=0.80, α=0.05, and β=0.20. Considering that the sample size may decrease due to different reasons in the study, it is planned to have a sample of 60 individuals, with 30 patients in each group.

Dependent and Independent Variables:

Independent variables: Socio-demographic characteristics of patients diagnosed with COPD (Age, gender, education, etc.), respiratory exercises (pursed-lip breathing exercise and diaphragmatic breathing exercise) Dependent variables: Vital signs (respiratory rate, SpO2 value, heart rate, blood pressure), 6-minute walk test, Modified Borg Scale score, Saint George Respiratory Questionnaire (Activity score) score, COPD sleep quality scale

Hypotheses:

H1: The application of respiratory exercises in COPD patients has a positive effect on reducing dyspnea severity.

H2: The application of respiratory exercises in COPD patients has a positive effect on activity level.

H3: The application of respiratory exercises in COPD patients has a positive effect on sleep quality.

Data Evaluation:

The SPSS program will be used for statistical analysis of the obtained data. Descriptive statistical analyses (number, percentage, mean, standard deviation) will be performed for the data. The Shapiro-Wilk test will be used to test whether the data show normal distribution. If the data show normal distribution, paired samples t-test and one-way ANOVA test will be used for matched sets. If the data do not show normal distribution, Kruskal Wallis and Wilcoxon tests will be used. Values with a p-value below 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and above
* Diagnosed with COPD for at least six months
* Modified Borg Dyspnea Scale score of at least 3
* Unable to complete the 6-minute walk test
* Not previously participated in a respiratory exercise program

Exclusion Criteria:

* Having cognitive impairment
* Not willing to participate in the study
* Failure to perform respiratory exercises regularly
* Having non-COPD lung diseases such as tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Modified Borg Scale(MBS) (for dyspnea severity of the COPD patients) | pre-intervention (first measurement)
  Dyspnea severity of the COPD patient will be evaluated with Modified Borg Scale(MBS). It was aimed to determine the change in dyspnea severity in COPD patients who received and regularly practiced video-based breathing exercises training. Modified Borg Scale (MBS): As scores increase, dyspnea severity increases (0: None, 0.5: Very, very light, 1: Very light, 2: Light, 3: Moderate, 4: Somewhat severe, 5: Severe, 6: ..., 7: Very severe, 8: ..., 9: Very, very severe, 10: Maximum).
St. George's respiratory questionnaire (for activity level of the COPD patients) | pre-intervention (first measurement)
  30 days of regular breathing exercise was aimed to realize the change in the activity level of patients with COPD. The change in activity level will be measured by Saint George's Respiratory Questionnaire (SGRQ). Saint George's Respiratory Questionnaire (SGRQ): The questionnaire consists of 50 items and three subscales: symptoms (8 items), activity (16 items), and impacts of the disease (26 items). Each item in the scale has an empirically determined weight. The questionnaire evaluates respiratory symptoms, activities limited by dyspnea, and the overall impact on daily life. Each subscale of the questionnaire is scored separately, and a total score is calculated. The total score ranges from 0 to 100, where a score of 0 indicates no impairment in quality of life, while a score of 100 indicates a progressive deterioration in quality of life.
Chronic Obstructive Pulmonary Disease and Asthma Sleep Impact Scale (for sleep qualty of the COPD patients) | pre-intervention (first measurement)
  30 days of regular breathing exercise was aimed to realize the change in the sleep qualty of patients with COPD. The Asthma COPD Sleep Scale is a Likert scale consisting of a total of 7 items. A high scale score indicates poor sleep quality and a low scale score indicates good sleep quality. In the scale, scores can range from a minimum of 0 to a maximum of 35. However, the original version of the scale does not specify minimum, maximum, or cut-off scores. A higher total score indicates poorer sleep quality, while a lower total score reflects better sleep quality. Relevant explanations regarding this matter are also provided.

SECONDARY OUTCOMES:
Modified Borg Scale(MBS) (for dyspnea severity of the COPD patients) | Last measurement 4 weeks after the first measurement (30 days later)
  Dyspnea severity of the COPD patient will be evaluated with Modified Borg Scale(MBS). It was aimed to determine the change in dyspnea severity in COPD patients who received and regularly practiced video-based breathing exercises training. Modified Borg Scale (MBS): As scores increase, dyspnea severity increases (0: None, 0.5: Very, very light, 1: Very light, 2: Light, 3: Moderate, 4: Somewhat severe, 5: Severe, 6: ..., 7: Very severe, 8: ..., 9: Very, very severe, 10: Maximum).
St. George's respiratory questionnaire (for activity level of the COPD patients) | Last measurement 4 weeks after the first measurement (30 days later)
  30 days of regular breathing exercise was aimed to realize the change in the activity level of patients with COPD. The change in activity level will be measured by Saint George's Respiratory Questionnaire (SGRQ). Saint George's Respiratory Questionnaire (SGRQ): The questionnaire consists of 50 items and three subscales: symptoms (8 items), activity (16 items), and impacts of the disease (26 items). Each item in the scale has an empirically determined weight. The questionnaire evaluates respiratory symptoms, activities limited by dyspnea, and the overall impact on daily life. Each subscale of the questionnaire is scored separately, and a total score is calculated. The total score ranges from 0 to 100, where a score of 0 indicates no impairment in quality of life, while a score of 100 indicates a progressive deterioration in quality of life.
Asthma Sleep Impact Scale (for sleep qualty of the COPD patients) | Last measurement 4 weeks after the first measurement (30 days later)
  30 days of regular breathing exercise was aimed to realize the change in the sleep qualty of patients with COPD. The Asthma COPD Sleep Scale is a Likert scale consisting of a total of 7 items. A high scale score indicates poor sleep quality and a low scale score indicates good sleep quality. In the scale, scores can range from a minimum of 0 to a maximum of 35. However, the original version of the scale does not specify minimum, maximum, or cut-off scores. A higher total score indicates poorer sleep quality, while a lower total score reflects better sleep quality. Relevant explanations regarding this matter are also provided.
  The effect of video-based breathing exercise training and regular practice on sleep quality will be measured with the same measurement tool (Asthma and Chronic Obstructive Pulmonary Disease Sleep Scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Bartin University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albarrati AM, Gale NS, Munnery MM, Cockcroft JR, Shale DJ. Daily physical activity and related risk factors in COPD. BMC Pulm Med. 2020 Mar 5;20(1):60. doi: 10.1186/s12890-020-1097-y. PMID 32138714
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Burkow TM, Vognild LK, Johnsen E, Bratvold A, Risberg MJ. Promoting exercise training and physical activity in daily life: a feasibility study of a virtual group intervention for behaviour change in COPD. BMC Med Inform Decis Mak. 2018 Dec 18;18(1):136. doi: 10.1186/s12911-018-0721-8. PMID 30563507
- [Background] Ceyhan Y, Tekinsoy Kartin P. The effects of breathing exercises and inhaler training in patients with COPD on the severity of dyspnea and life quality: a randomized controlled trial. Trials. 2022 Aug 26;23(1):707. doi: 10.1186/s13063-022-06603-3. PMID 36028881
- [Background] Chang CH, Chuang LP, Lin SW, Lee CS, Tsai YH, Wei YF, Cheng SL, Hsu JY, Kuo PH, Yu CJ, Chen NH. Factors responsible for poor sleep quality in patients with chronic obstructive pulmonary disease. BMC Pulm Med. 2016 Aug 8;16(1):118. doi: 10.1186/s12890-016-0281-6. PMID 27501837
- [Background] de Roos P, Lucas C, Strijbos JH, van Trijffel E. Effectiveness of a combined exercise training and home-based walking programme on physical activity compared with standard medical care in moderate COPD: a randomised controlled trial. Physiotherapy. 2018 Mar;104(1):116-121. doi: 10.1016/j.physio.2016.08.005. Epub 2017 Jul 14. PMID 28802772
- [Background] Hanania NA, O'Donnell DE. Activity-related dyspnea in chronic obstructive pulmonary disease: physical and psychological consequences, unmet needs, and future directions. Int J Chron Obstruct Pulmon Dis. 2019 May 24;14:1127-1138. doi: 10.2147/COPD.S188141. eCollection 2019. PMID 31213793
- [Background] Jones PW. Health status measurement in chronic obstructive pulmonary disease. Thorax. 2001 Nov;56(11):880-7. doi: 10.1136/thorax.56.11.880. PMID 11641515
- [Background] Ko FW, Tam W, Siu EHS, Chan KP, Ngai JC, Ng SS, Chan TO, Hui DS. Effect of short-course exercise training on the frequency of exacerbations and physical activity in patients with COPD: A randomized controlled trial. Respirology. 2021 Jan;26(1):72-79. doi: 10.1111/resp.13872. Epub 2020 Jun 15. PMID 32542906
- [Background] Ierodiakonou D, Bouloukaki I, Kampouraki M, Papadokostakis P, Poulorinakis I, Lampraki I, Athanasiou P, Schiza S, Tsiligianni I; Greek UNLOCK Group. Subjective sleep quality is associated with disease status in COPD patients. The cross-sectional Greek UNLOCK study. Sleep Breath. 2020 Dec;24(4):1599-1605. doi: 10.1007/s11325-020-02039-8. Epub 2020 Feb 26. PMID 32103395
- [Background] Lewthwaite H, Effing TW, Olds T, Williams MT. Physical activity, sedentary behaviour and sleep in COPD guidelines: A systematic review. Chron Respir Dis. 2017 Aug;14(3):231-244. doi: 10.1177/1479972316687224. Epub 2017 Feb 24. PMID 28774202
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Mayer AF, Karloh M, Dos Santos K, de Araujo CLP, Gulart AA. Effects of acute use of pursed-lips breathing during exercise in patients with COPD: a systematic review and meta-analysis. Physiotherapy. 2018 Mar;104(1):9-17. doi: 10.1016/j.physio.2017.08.007. Epub 2017 Aug 31. PMID 28969859
- [Background] McNicholas WT, Hansson D, Schiza S, Grote L. Sleep in chronic respiratory disease: COPD and hypoventilation disorders. Eur Respir Rev. 2019 Sep 25;28(153):190064. doi: 10.1183/16000617.0064-2019. Print 2019 Sep 30. PMID 31554703
- [Background] Ozer Z, Bahcecioglu Turan G, Aksoy M. The effects of yoga on dyspnea, sleep and fatigue in chronic respiratory diseases. Complement Ther Clin Pract. 2021 May;43:101306. doi: 10.1016/j.ctcp.2021.101306. Epub 2021 Jan 19. PMID 33545575
- [Background] Pokrzywinski RF, Meads DM, McKenna SP, Glendenning GA, Revicki DA. Development and psychometric assessment of the COPD and Asthma Sleep Impact Scale (CASIS). Health Qual Life Outcomes. 2009 Dec 7;7:98. doi: 10.1186/1477-7525-7-98. PMID 19968881
- [Background] Polat H, Erguney S. The Effect of Reflexology Applied to Patients with Chronic Obstructive Pulmonary Disease on Dyspnea and Fatigue. Rehabil Nurs. 2017 Jan/Feb;42(1):14-21. doi: 10.1002/rnj.266. PMID 26956942
- [Background] Rennard S, Decramer M, Calverley PM, Pride NB, Soriano JB, Vermeire PA, Vestbo J. Impact of COPD in North America and Europe in 2000: subjects' perspective of Confronting COPD International Survey. Eur Respir J. 2002 Oct;20(4):799-805. doi: 10.1183/09031936.02.03242002. PMID 12412667
- [Background] Rossi RC, Vanderlei FM, Bernardo AF, Souza NM, Goncalves AC, Ramos EM, Pastre CM, Abreu LC, Vanderlei LC. Effect of pursed-lip breathing in patients with COPD: Linear and nonlinear analysis of cardiac autonomic modulation. COPD. 2014 Feb;11(1):39-45. doi: 10.3109/15412555.2013.825593. Epub 2013 Oct 10. PMID 24111515
- [Background] Serin EK, Ister ED, Ozdemir A. The relationship between sleep quality and dyspnoea severity in patients with COPD. Afr Health Sci. 2020 Dec;20(4):1785-1792. doi: 10.4314/ahs.v20i4.32. PMID 34394240
- [Background] Seyedi Chegeni P, Gholami M, Azargoon A, Hossein Pour AH, Birjandi M, Norollahi H. The effect of progressive muscle relaxation on the management of fatigue and quality of sleep in patients with chronic obstructive pulmonary disease: A randomized controlled clinical trial. Complement Ther Clin Pract. 2018 May;31:64-70. doi: 10.1016/j.ctcp.2018.01.010. Epub 2018 Feb 6. PMID 29705482
- [Background] Ubolnuar N, Tantisuwat A, Thaveeratitham P, Lertmaharit S, Kruapanich C, Chimpalee J, Mathiyakom W. Effects of pursed-lip breathing and forward trunk lean postures on total and compartmental lung volumes and ventilation in patients with mild to moderate chronic obstructive pulmonary disease: An observational study. Medicine (Baltimore). 2020 Dec 18;99(51):e23646. doi: 10.1097/MD.0000000000023646. PMID 33371099
- [Background] Vukoja M, Kopitovic I, Milicic D, Maksimovic O, Pavlovic-Popovic Z, Ilic M. Sleep quality and daytime sleepiness in patients with COPD and asthma. Clin Respir J. 2018 Feb;12(2):398-403. doi: 10.1111/crj.12528. Epub 2016 Jul 27. PMID 27402309
- [Background] Yang Y, Wei L, Wang S, Ke L, Zhao H, Mao J, Li J, Mao Z. The effects of pursed lip breathing combined with diaphragmatic breathing on pulmonary function and exercise capacity in patients with COPD: a systematic review and meta-analysis. Physiother Theory Pract. 2022 Jul;38(7):847-857. doi: 10.1080/09593985.2020.1805834. Epub 2020 Aug 18. PMID 32808571
- [Background] Yilmaz CK, Kapucu S. The Effect of Progressive Relaxation Exercises on Fatigue and Sleep Quality in Individuals With COPD. Holist Nurs Pract. 2017 Nov/Dec;31(6):369-377. doi: 10.1097/HNP.0000000000000234. PMID 29028775